CLINICAL TRIAL: NCT04424407
Title: A Novel Use of a Sleep Intervention to Target the Emotion Regulation Brain Network to Treat Depression and Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Goldstein-Piekarski, Assistant Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-56961; R61MH120245 (NIH)
Record Dates: First submitted 2020-06-03; First posted 2020-06-11 (Actual); Results first posted 2025-10-15 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-09

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Anxiety; CBT-I; Cognitive Behavioral Therapy for Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This is a single-armed trial. All participants will receive Cognitive Behavioral Therapy for Insomnia
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT-I (Other)
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Participants will meet with a psychologist once a week for six weeks to complete a brief CBT-I intervention. Cognitive Behavioral Therapy for Insomnia consists of a cognitive therapy and a behavioral therapy. The cognitive therapy is designed to identify incorrect ideas about sleep, challenge their validity, and replace them with correct information. This therapy tries to reduce worry, anxiety, and fear that one won't sleep by providing accurate information about sleep. The behavioral therapy increases sleep quality by limiting excessive time spent in bed to increase homeostatic sleep drive and sleep consolidation.
  Other Names: CBT-I

SUMMARY:
Several lines of evidence suggest that unhealthy sleep patterns contribute to depressive symptoms through disruption of brain networks that regulate emotional functions. However, we do not yet know to what degree the emotion regulation brain network is modified by the restoration of sleep, or whether the degree to which a sleep intervention modifies these neural targets mediates reductions in other depressive symptoms including suicidality.

The overall aim is to test the efficacy of an established sleep intervention (Cognitive Behavioral Therapy for Insomnia (CBT-I)) in reducing depressive symptoms through improving emotion regulation brain function in individuals with elevated depressive symptoms and clinically meaningful sleep disturbance.

In this study, we will assess feasibility of recruitment and retention as well as target engagement. Target engagement is defined as the treatment effect on increasing mPFC-amygdala connectivity, and/or decreasing amygdala reactivity during emotion reactivity and regulation paradigms. Participants will be 70 adults experiencing at least moderate sleep disturbances and who also have elevated anxious and/or depressive symptoms. Emotion distress and sleep disruption will be assessed prior to, and weekly while receiving six Cognitive Behavioral Therapy for Insomnia (CBT-I) across a period of 8 weeks. CBT-I improves sleep patterns through a combination of sleep restriction, stimulus control, mindfulness training, cognitive therapy targeting dysfunctional beliefs about sleep, and sleep hygiene education. Using fMRI scanning, emotion regulation network neural targets will be assayed prior to and following completion of CBT-I treatment.

ELIGIBILITY:
Inclusion Criteria:

* Ages 25-60
* Subjective complaint of sleep disturbance for ≥ 3 months (ISI≥10)
* Subjective complaint of depression (BDI≥14) and not at imminent risk for suicide, as measured by CSSRS assessment
* Fluent and literate in English
* Written informed consent.
* Reside within 60 miles of Stanford University

Exclusion Criteria:

* Presence of other sleep or circadian rhythm disorders
* Medications that would significantly impact sleep, alertness, or mood
* >14 alcoholic drinks per week or >4 drinks per occasion
* General medical condition, disease or neurological disorder that interferes with the assessments or outpatient participation
* Substance abuse or dependence
* Mild traumatic brain injury
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to follow study protocols
* Pregnant or breast feeding
* Current or lifetime history of bipolar disorder or psychosis
* Current or or expected cognitive behavior therapy or other evidence-based psychotherapies for another condition
* Received CBT-I within the past year
* Acute or unstable chronic illness
* Current exposure to trauma, or exposure to trauma within the past 3 months
* Working a rotating shift that overlaps with 2400h.
* Presence of suicidal ideations representing imminent risk as determined by the empirically-supported, standardized suicide risk assessment" to the exclusion criteria
* Individuals who are not CPAP adherent or have untreated OSA of moderate severity or worse (AHI ≥ 15)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2024-03-23 (Actual); Study Completion 2024-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Goldstein-Piekarski, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- CBT-I: Cognitive Behavioral Therapy (CBT) for Insomnia: Participants will meet with a psychologist once a week for six weeks to complete a brief CBT-I intervention. Cognitive Behavioral Therapy for Insomnia consists of a cognitive therapy and a behavioral therapy. The cognitive therapy is designed to identify incorrect ideas about sleep, challenge their validity, and replace them with correct information. This therapy tries to reduce worry, anxiety, and fear that one won't sleep by providing accurate information about sleep. The behavioral therapy increases sleep quality by limiting excessive time spent in bed to increase homeostatic sleep drive and sleep consolidation.
Period: Overall Study
Arm/Group | CBT-I
Started | 51
Completed | 48
Not Completed | 3
Not completed — Withdrawal by Subject | 2
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | CBT-I
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.2 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 51
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 18
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 28
  More than one race | 2
  Unknown or Not Reported | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Amygdala Activation During the Facial Expressions of Emotion Task (Conscious Condition) as Assessed by Functional Magnetic Resonance Imaging
Description: The Conscious condition of the Facial Expressions of Emotion task measures supraliminal (without backward masking) emotional face processing. Amygdala activation while viewing threat-related emotional faces relative to neutral faces was quantified using functional magnetic resonance imaging (fMRI) as a marker of Emotion Regulation Network engagement. Blood-oxygenation level dependent (BOLD) signal change before and after CBT-I treatment was compared by modeling the activity of the amygdala while viewing emotional faces using generalized linear models, producing beta weights for each participant and timepoint. A positive beta-weight at pre-treatment means that the amygdala increased its activity in response to emotional faces, relative to neutral faces. A negative value for the change in amygdala activation means that average amygdala reactivity decreased following treatment. It is theorized that higher amygdala emotional reactivity is associated with worse outcomes.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed the pre-treatment baseline, and who had interpretable image data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Beta weights (arbitrary units)
Groups:
- Pre-treatment Amygdala Activation: Baseline amygdala activation before CBT-I treatment.
- Change in Amygdala Activation: Post-treatment amygdala reactivity minus pre-treatment amygdala reactivity.
Arm/Group | Pre-treatment Amygdala Activation | Change in Amygdala Activation
Number analyzed (Participants) | 44 | 41
Beta weights (arbitrary units)
  Fear > Neutral | 0.11 (0.32) | -0.18 (0.34)
  Threat > Neutral | 0.22 (0.60) | -0.25 (0.63)
  Anger > Neutral | 0.11 (0.36) | -0.07 (0.40)
Statistical Analysis 1: Comparison: Change in Amygdala Activation; Analysis of Conscious Fear > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.008, Mixed Models Analysis — P-values from linear mixed effects models were False Discovery Rate-adjusted (Benjamini-Hochberg method) for the number of contrasts (3) in the Conscious Faces task. The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Change in Amygdala Activation; Analysis of Conscious Threat > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.08, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: Change in Amygdala Activation; Analysis of Conscious Anger > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.49, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]

2. Primary Outcome: Change in Amygdala Activation During the Facial Expressions of Emotion Task (Nonconscious Condition) as Assessed by Functional Magnetic Resonance Imaging
Description: The Nonconscious condition of the Facial Expressions of Emotion task measures subliminal (with backward masking) emotional face processing. Amygdala activation while viewing threat-related emotional faces relative to neutral faces was quantified using fMRI as a marker of Emotion Regulation Network engagement. Blood-oxygenation level dependent (BOLD) signal change before and after CBT-I treatment was compared by modeling the activity of the amygdala while viewing emotional faces using generalized linear models, producing beta weights for each participant and timepoint. A positive beta-weight at pre-treatment means that the amygdala increased its activity in response to emotional faces, relative to neutral faces. A negative value for the change in amygdala activation means that average amygdala reactivity decreased following treatment. It is theorized that higher amygdala emotional reactivity is associated with worse outcomes.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable image data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Beta weights (arbitrary units)
Groups:
- Change in Amygdala Activaiton: Post-treatment amygdala reactivity minus pre-treatment amygdala reactivity.
Arm/Group | Pre-treatment Amygdala Activation | Change in Amygdala Activaiton
Number analyzed (Participants) | 46 | 44
Beta weights (arbitrary units)
  Fear > Neutral | -0.01 (0.24) | -0.01 (0.35)
  Threat > Neutral | 0.009 (0.41) | -0.01 (0.58)
  Anger > Neutral | 0.02 (0.22) | 0.001 (0.30)
Statistical Analysis 1: Comparison: Change in Amygdala Activaiton; Analysis of Nonconscious Fear > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.99, Mixed Models Analysis — P-values from linear mixed effects models were False Discovery Rate-adjusted (Benjamini-Hochberg method) for the number of contrasts (3) in the Nonconscious Faces task. The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Change in Amygdala Activaiton; Analysis of Nonconscious Threat > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.99, Mixed Models Analysis — [p-value comment as in outcome 2, analysis 1]

3. Primary Outcome: Change in Amygdala Activation During the Emotion Regulation Scenes Task
Description: Participants are asked to "look" or "decrease" their emotional response to negative and neutral valence images taken from the International Affective Picture System. Amygdala activation while viewing emotional scenes relative to neutral scenes, and while passively viewing emotional scenes relative to down-regulating emotion, was quantified using fMRI as a marker of Emotion Regulation Network engagement. Blood-oxygenation level dependent (BOLD) signal change before and after CBT-I treatment was compared by modeling the activity of the amygdala while viewing emotional scenes or while downregulating using generalized linear models, producing beta weights for each participant and timepoint. A positive beta-weight at pre-treatment means that the amygdala increased its activity in response to the task demands, and a negative value means that average amygdala reactivity decreased following treatment. It is theorized that higher amygdala emotional reactivity is associated with worse outcomes
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable image data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Beta weights (arbitrary units)
Arm/Group | Pre-treatment Amygdala Activation | Change in Amygdala Activation
Number analyzed (Participants) | 44 | 42
Beta weights (arbitrary units)
  Negative > Neutral | 0.35 (0.56) | 0.05 (0.71)
  Look Negative > Decrease Negative | -0.05 (0.28) | 0.03 (0.39)
Statistical Analysis 1: Comparison: Change in Amygdala Activation; Analysis of Emotion Regulation Scenes task Negative > Neutral amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.65, Mixed Models Analysis — P-values from linear mixed effects models were False Discovery Rate-adjusted (Benjamini-Hochberg method) for the number of contrasts (2) in the Emotion Regulation Scenes task. The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Change in Amygdala Activation; Analysis of Emotion Regulation Scenes task Look Negative > Decrease Negative amygdala reactivity was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.65, Mixed Models Analysis — [p-value comment as in outcome 3, analysis 1]

4. Primary Outcome: Change in Amygdala-Medial Prefrontal Cortex Connectivity During the Facial Expressions of Emotion Task (Conscious Condition) as Assessed by Functional Magnetic Resonance Imaging
Description: This outcome tested whether amygdala connectivity with regions of the mPFC was changed following treatment using psychophysiological interaction (PPI) analysis for this contrast/task. Regions of the mPFC include: dorsal anterior cingulate cortex (dACC), ventromedial prefrontal cortex (vmPFC), dorsomedial prefrontal cortex (dmPFC), subgenual anterior cingulate cortex (sgACC), pregenual anterior cingulate cortex (pACC). PPI analyses produce a beta weight for each participant at each timepoint, and represents the degree to which the connectivity of the amygdala and mPFC is modulated by task conditions. A positive value means average connectivity increases in the task-contrast, and a positive value for the change score means an increase in average connectivity following CBT-I treatment. It is theorized that higher amygdala connectivity is associated with better outcomes.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable image data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Beta weights (arbitrary units)
Groups:
- Pre-treatment Amygdala-mPFC Connectivity: Baseline amygdala-mPFC connectivity before CBT-I treatment.
- Change in Amygdala-mPFC Connectivity: Amygdala-mPFC connectivity at Post-treatment minus pre-treatment.
Arm/Group | Pre-treatment Amygdala-mPFC Connectivity | Change in Amygdala-mPFC Connectivity
Number analyzed (Participants) | 44 | 41
Beta weights (arbitrary units)
  Amygdala-dACC Connectivity | 0.004 (0.49) | 0.02 (0.63)
  Amygdala-dmPFC Connectivity | -0.04 (0.46) | -0.02 (0.66)
  Amygdala-pACC Connectivity | 0.007 (0.55) | -0.10 (0.60)
  Amygdala-sgACC Connectivity | -0.09 (0.39) | 0.14 (0.49)
  Amygdala-vmPFC Connectivity | -0.08 (0.51) | -0.10 (0.55)
Statistical Analysis 1: Comparison: Change in Amygdala-mPFC Connectivity; Analysis of amygdala-dACC connectivity from the Conscious Fear > Neutral task/contrast was done by applying linear mixed effects models testing the effect of treatment-time on connectivity. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.86, Mixed Models Analysis — P-values from linear mixed effects models were False Discovery Rate-adjusted (Benjamini-Hochberg method) for the number of mPFC regions (5). The a priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Change in Amygdala-mPFC Connectivity; Analysis of amygdala-dmPFC connectivity from the Conscious Fear > Neutral task/contrast was done by applying linear mixed effects models testing the effect of treatment-time on connectivity. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.86, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Change in Amygdala-mPFC Connectivity; Analysis of amygdala-pACC connectivity from the Conscious Fear > Neutral task/contrast was done by applying linear mixed effects models testing the effect of treatment-time on connectivity. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.83, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Change in Amygdala-mPFC Connectivity; Analysis of amygdala-sgACC connectivity from the Conscious Fear > Neutral task/contrast was done by applying linear mixed effects models testing the effect of treatment-time on connectivity. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.23, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Change in Amygdala-mPFC Connectivity; Analysis of amygdala-vmPFC connectivity from the Conscious Fear > Neutral task/contrast was done by applying linear mixed effects models testing the effect of treatment-time on connectivity. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.83, Mixed Models Analysis — [p-value comment as in outcome 4, analysis 1]

5. Primary Outcome: Change in Beck Depression Inventory (BDI)
Description: This measure is of the Beck Depression Inventory-II total score after excluding one sleep item.
  The BDI-II is a 21-item self-report scale with high validity and reliability that assesses the severity of depression symptoms. The depression items consist of: sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, and loss of interest in sex. Items are scored from 0 to 3, and summed to create an overall score of 0 to 63. higher scores indicate greater levels of severity. The ranges for depression are: 0-13 minimal, 14-19 mild, 20-28 moderate, and 29-63 severe. A negative change score means that average depression symptom severity was reduced following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: All participants who competed pre-treatment baseline and with interpretable data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-treatment: Depression symptom severity prior to CBT-I
- Change in Depression Symptom Severity: Post-treatment depression symptom severity score minus pre-treatment depression symptom severity score.
Arm/Group | Pre-treatment | Change in Depression Symptom Severity
Number analyzed (Participants) | 47 | 47
units on a scale | 17.5 (6.2) | -6.61 (7.6)
Statistical Analysis 1: Comparison: Change in Depression Symptom Severity; Analysis of change in depression symptom severity score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p < 0.0001, Mixed Models Analysis — P-values are from linear mixed effects models. The a priori threshold for statistical significance was < 0.05

6. Primary Outcome: Change in PSG Sleep Efficiency
Description: Sleep efficiency (SE) is the percentage of total time in bed actually spent sleeping. Based on the overnight PSG sleep recording, SE will be calculated as the total time (minutes) spent asleep (sum of Stages N1, N2, N3, and REM) divided by the total time (minutes) in bed, and multiplied by 100. A positive change score means average sleep efficiency increased following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable image data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Sleep Efficiency (%)
Groups:
- Pre-treatment: PSG Sleep efficiency prior to CBT-I treatment.
- Change in PSG Sleep Efficiency: Post-treatment sleep efficiency minus pre-treatment sleep efficiency.
Arm/Group | Pre-treatment | Change in PSG Sleep Efficiency
Number analyzed (Participants) | 45 | 42
Sleep Efficiency (%) | 78.9 (15.1) | 8.57 (15.56)
Statistical Analysis 1: Comparison: Change in PSG Sleep Efficiency; Analysis of change in sleep efficiency was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.002, Mixed Models Analysis — P-values are from linear mixed effects models. The a priori threshold for statistical significance was < 0.05

7. Secondary Outcome: Change in Beck Scale of Suicidal Ideation Total Score
Description: The Beck Scale of Suicidal Ideation (BSSI) is designed to assess the severity of suicidal ideation over the past week. The total score is derived from the sum of the first 19 items, creating an overall score ranging from 0 to 38. Scores of 0 are interpreted as no suicidal ideation, 1-8 as low levels, 9-16 as moderate levels, and 17-38 as high levels. A negative change score means an average reduction in suicidal ideation following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Pre-treatment: Suicidal thinking prior to CBT-I treatment.
- Change in Suicidal Thinking: Post-treatment suicidal thinking minus pre-treatment suicidal thinking.
Arm/Group | Pre-treatment | Change in Suicidal Thinking
Number analyzed (Participants) | 47 | 47
score on a scale | 1.74 (3.88) | -1.11 (4.80)
Statistical Analysis 1: Comparison: Change in Suicidal Thinking; Analysis of change in suicidal ideation score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p < 0.0001, Mixed Models Analysis — P-values are from linear mixed effects models. The a priori threshold for statistical significance was < 0.05

8. Secondary Outcome: Change in Columbia Suicide Severity Rating Scale
Description: The Columbia Suicide Severity Rating Scale (CSSRS) is a 12-item checklist that was designed to quantify the severity of suicidal ideation and behavior. It is composed of two parts. The first six questions ask about suicidal ideation and behavior in the past month while the last six questions ask about suicidal ideation and behavior since the last visit. The CSSRS has been proven to be reliable and valid. It has also been shown to have high sensitivity and specificity to the different suicidal behavior classifications. The CSSRS does not provide a numerical score but categorizes risk levels based on responses. We report the proportions of risk at each timepoint.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable CSSRS data at the respective timepoint.
Measure: Count of Participants; unit: Participants
Groups:
- Pre-treatment: Suicidal thinking before CBT-I treatment.
- Post-treatment: Suicidal thinking following CBT-I treatment.
Arm/Group | Pre-treatment | Post-treatment
Number analyzed (Participants) | 50 | 47
Participants
  No Risk | 37 | 41
  Low Risk | 13 | 5
  Moderate Risk | 0 | 1
  High Risk | 0 | 0
Statistical Analysis 1: Comparison: Pre-treatment vs Post-treatment; Analysis of change in suicidal risk was done by applying ordinal logistic regression (proportional odds model) testing the effect of treatment-time on the probability of being in a higher risk category. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.03, Mixed Models Analysis — P-values are uncorrected from ordinal logistic regression model. The a priori threshold for statistical significance was < 0.05; A significant p-value here means that treatment was associated with reduced odds of being in a higher risk category

9. Secondary Outcome: Change in Actigraph Sleep Onset Latency (SOL) as a Measure of Sleep Continuity
Description: Sleep Onset Latency (SOL) is the time (minutes) from "lights out" to actually falling asleep (sleep onset).
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

10. Secondary Outcome: Change in Actigraph Number of Arousals as a Measure of Sleep Continuity
Description: Number of Arousals is determined by number of times of awakening as seen on the actigraph data.
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

11. Secondary Outcome: Change in Actigraph Wake After Sleep Onset (WASO) as a Measure of Sleep Continuity
Description: Wake After Sleep Onset (WASO) are periods of wakefulness occurring after sleep onset, before final awakening (sleep offset).
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

12. Secondary Outcome: Change in Actigraph Total Sleep Time (TST) as a Measure of Sleep Continuity
Description: Total Sleep Time (TST) is the total time spent asleep, from the start of sleep onset to sleep offset subtracting any periods of wakefulness.
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

13. Secondary Outcome: Change in Actigraph Sleep Efficiency (SE) as a Measure of Sleep Continuity
Description: Sleep Efficiency (SE) is calculated as TST divided by total time spent in bed, multiplied by 100.
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

14. Secondary Outcome: Change in PSG Sleep Onset Latency (SOL) as a Measure of Sleep Architecture
Description: Sleep onset latency is the time it takes to fall asleep, specifically the amount of time in minutes from "LightsOff", which is the time at which the participant started trying to sleep, to stage 1 sleep. A negative change score means it took less time to fall asleep following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable PSG data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Pre-treatment: Sleep onset latency prior to CBT-I treatment.
- Change in PSG Sleep Onset Latency: Sleep onset latency (PSG) following CBT-I treatment.
Arm/Group | Pre-treatment | Change in PSG Sleep Onset Latency
Number analyzed (Participants) | 36 | 33
Minutes | 30.29 (39.34) | -11.44 (47.96)
Statistical Analysis 1: Comparison: Change in PSG Sleep Onset Latency; Analysis of change in sleep onset latency (PSG) was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.28, Mixed Models Analysis

15. Secondary Outcome: Change in PSG Number of Arousals as a Measure of Sleep Architecture
Description: Number of Arousals is determined by number of times of awakening by EEG changes. A negative change score means on average there were fewer overnight arousals following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable PSG data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Number of Awakenings
Groups:
- Pre-treatment: Number of arousals before CBT-I treatment.
- Change in Number of Arousals: Post-treatment number of arousals minus pre-treatment number of arousals
Arm/Group | Pre-treatment | Change in Number of Arousals
Number analyzed (Participants) | 45 | 42
Number of Awakenings | 21.96 (7.3) | -1.44 (9.67)
Statistical Analysis 1: Comparison: Change in Number of Arousals; Analysis of change in number of awakenings derived from PSG was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.33, Mixed Models Analysis — P-values are uncorrected from linear mixed effects models. The a priori threshold for statistical significance was < 0.05

16. Secondary Outcome: Change in PSG Wake After Sleep Onset (WASO) as a Measure of Sleep Architecture
Description: Wake After Sleep Onset (WASO) are periods of wakefulness occurring after sleep onset, before final awakening (sleep offset) measured by EEG changes. A negative change value means there was less WASO on average after CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable PSG data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Pre-treatment: PSG WASO before CBT-I treatment.
- Change in PSG WASO: Post-treatment PSG WASO minus pre-treatment WASO
Arm/Group | Pre-treatment | Change in PSG WASO
Number analyzed (Participants) | 45 | 42
Minutes | 58.3 (63.02) | -27.74 (66.42)
Statistical Analysis 1: Comparison: Change in PSG WASO; Analysis of change in wake after sleep onset (WASO) was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.013, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

17. Secondary Outcome: Change in PSG Total Sleep Time (TST) as a Measure of Sleep Architecture
Description: Total Sleep Time (TST) is the total time (minutes) spent asleep, from the start of sleep onset to sleep offset, subtracting any periods of wakefulness. TST includes stages N1, N2, N3, and REM sleep. A positive change score means the average TST increased following CBT-I.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had interpretable PSG data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Minutes
Groups:
- Pre-treatment: TST before CBT-I treatment.
- Change in PSG TST: Post-treatment PSG TST minus Pre-treatment PSG TST
Arm/Group | Pre-treatment | Change in PSG TST
Number analyzed (Participants) | 45 | 42
Minutes | 362.23 (93.31) | 5.67 (103.27)
Statistical Analysis 1: Comparison: Change in PSG TST; Analysis of change in PSG TST was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.66, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

18. Secondary Outcome: Change in Sleep Physiology Measured by PSG
Description: Fronto-central EEG power spectral density analysis associated with sleep stages will be calculated in the Delta (0.5-Hz), Theta (4-7Hz), Alpha (7-11Hz), Sigma (12-15Hz), Beta-1 (15-20Hz), Beta-2 (20-35Hz) and Gamma (35-45Hz) bands, according to published methods. A positive change score means there was an increase in absolute power in the specified frequency band following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: All participants who competed pre-treatment baseline and with interpretable PSG data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: Absolute spectral power, µV²/Hz
Groups:
- Pre-treatment: Spectral EEG power before CBT-I treatment.
- Change in Spectral EEG Power: Post-treatment power minus pre-treatment power.
Arm/Group | Pre-treatment | Change in Spectral EEG Power
Number analyzed (Participants) | 28 | 33
Absolute spectral power, µV²/Hz
  Delta (0.5-4Hz) | 29.52 (2.41) | 0.04 (1.56)
  Theta (4-7Hz) | 18.77 (2.29) | 0.40 (1.40)
  Alpha (7-11Hz) | 17.47 (2.68) | 0.37 (1.03)
  Sigma (12-15Hz) | 14.03 (2.85) | 0.25 (1.23)
  Beta-1 (15-20Hz) | 9.82 (2.68) | 0.15 (1.11)
  Beta-2 (20-35Hz) | 9.23 (2.36) | 0.08 (1.29)
  Gamma (35-45Hz) | 2.90 (1.86) | 0.13 (1.68)
Statistical Analysis 1: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Delta absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.96, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Theta absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.23, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 3: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Alpha absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.11, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 4: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Sigma absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.44, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 5: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Beta-1 absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.68, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 6: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Beta-2 absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.74, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 7: Comparison: Change in Spectral EEG Power; Analysis of change in PSG Gamma absolute power was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.84, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

19. Secondary Outcome: Change in Insomnia Severity Index (ISI) Scale Score
Description: Subjective ratings of sleep disturbance and insomnia severity will be assessed with the Insomnia Severity Index. The Insomnia Severity Index (ISI) is a 7-item self-report measure of insomnia type, severity, and impact on functioning. The items consist of severity of sleep onset, sleep maintenance, early morning awakenings, sleep dissatisfaction, interference with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Items are scored from 0 to 4 (0 = no problem, 4 = very severe problem), then summed to create an overall score of 0 to 28. Score ranges of insomnia are: 0-7 absent, 8-14 sub-threshold, 15-21 moderate, and 22-28 severe. The ISI has good validity and reliability. A negative change score means average insomnia symptoms improved following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed pre-treatment baseline, and who had ISI data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-treatment: Insomnia symptom severity before CBT-I treatment.
- Change in Insomnia Symptom Severity: Post-treatment insomnia symptom severity minus pre-treatment insomnia symptom severity.
Arm/Group | Pre-treatment | Change in Insomnia Symptom Severity
Number analyzed (Participants) | 48 | 47
units on a scale | 15.7 (3.83) | -7.98 (3.96)
Statistical Analysis 1: Comparison: Change in Insomnia Symptom Severity; Analysis of change in insomnia symptom severity score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

20. Secondary Outcome: Change in 36-Item Short Form Survey (SF-36) Score
Description: The SF-36 measures health-related quality of life based on eight domains: physical activity, social activities, limitations in activities due to physical health problems, bodily pain, general mental health, limitations in activities due to emotional problems, vitality, and general health perceptions. Items are recoded then averaged together to create each an average score for all items that the respondent answered. The eight subscales are then into two component summary t-scores (Mental and Physical Component Summary t-scores), each with a mean of 50 and a standard deviation of 10. A t-score higher than 50 means better mental or physical health than the general population, and a t-score below 50 means worse than the general population. Instructions for scoring these component scores recommends that they be set to missing if any subscales are missing. A positive change score means the Component Summary Score improved following CBT-I.
Time Frame: Assessed at week 0 and week 11
Population: Participants who completed the pre-treatment baseline, and who had interpretable SF-36 data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: t-score
Groups:
- Pre-treatment: Mental Component Summary and Physical Component Summary scores prior to CBT-I treatment.
- Change in Component Summary Scores: Post-treatment Mental Component Summary and Physical Component Summary scores minus pre-treatment scores.
Arm/Group | Pre-treatment | Change in Component Summary Scores
Number analyzed (Participants) | 50 | 47
t-score
  Mental Component T-Score | 31.72 (9.27) | 7.64 (14.59)
  Physical Component T-Score | 54.38 (6.75) | 0.25 (9.20)
Statistical Analysis 1: Comparison: Change in Component Summary Scores; Analysis of change in SF-36 Mental Component Score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]
Statistical Analysis 2: Comparison: Change in Component Summary Scores; Analysis of change in SF-36 Physical Component Score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p = 0.94, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

21. Secondary Outcome: Change in Beck Anxiety Inventory (BAI)
Description: The BAI is a 21-item self-report scale that assesses the severity of anxiety symptoms.
  Items are scored from 0 to 3 (0 = not at all, 3 = severe), then summed to create an overall score range of 0 to 63. Higher scores indicate greater levels of severity, and the ranges for anxiety levels are: 0-9 normal to minimal, 10-18 mild to moderate, 19-29 moderate to severe, and 30-63 severe. The BAI consists of two factors: somatic and cognitive. A negative change score means that average anxiety symptom severity was reduced following CBT-I treatment.
Time Frame: Assessed at week 0 and week 11
Population: All participants who competed pre-treatment baseline and with data at the respective timepoint.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Pre-treatment: Anxiety symptoms before CBT-I treatment.
- Change in Anxiety Symptom Severity: Post-treatment anxiety symptom severity score minus pre-treatment anxiety symptom severity score.
Arm/Group | Pre-treatment | Change in Anxiety Symptom Severity
Number analyzed (Participants) | 47 | 47
units on a scale | 9.87 (5.88) | -3.78 (7.97)
Statistical Analysis 1: Comparison: Change in Anxiety Symptom Severity; Analysis of change in anxiety symptom severity score was done by applying linear mixed effects models testing the effect of treatment-time. Random intercepts at the individual participant level are included to account for the clustering of observations within individuals across time. All statistical models include age and sex as covariates of non-interest; Test type: Other; p < 0.0001, Mixed Models Analysis — [p-value comment as in outcome 15, analysis 1]

22. Secondary Outcome: Change in Respiratory Sinus Arrhythmia (RSA)- Measured by PSG
Description: RSA is the phenomenon of an increased heart rate during inhalation and a decreased heart rate during exhalation. Since these fluctuations are controlled mainly by vagal influences on the heart, RSA serves as a reliable metric for measuring parasympathetic activity. RSA has been proven to be a reliable measure of emotion regulation and emotional responding in numerous studies.
Time Frame: Assessed at week 0 and week 11
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 11 weeks
Arm/Group | CBT-I
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 14/51
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT-I (N=51)
Mood Changes (Psychiatric disorders) | 8 (10)
Increased Anxiety (Psychiatric disorders) | 3 (3)
Fever/Cold Symptoms (Infections and infestations) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Original (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/07/NCT04424407/Prot_SAP_001.pdf
  • Statistical Analysis Plan: Revised (2025-05-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT04424407/SAP_002.pdf
  • Informed Consent Form (2023-08-18): https://cdn.clinicaltrials.gov/large-docs/07/NCT04424407/ICF_000.pdf